CLINICAL TRIAL: NCT03489603
Title: Valutazione Clinica e Farmacoeconomica Delle Metodiche di Dosaggio Per la TROponina CARdiaca Per la Diagnosi di NSTEMI Nel Setting Della Pratica Clinica Della Medicina di Pronto Soccorso Nel Territorio Nazionale
Brief Title: Clinical and Economic Outcomes of High Sensitivity Troponin for no ST Elevation Myocardial Infarction in Patients With Chest Pain in Emergency Departments in Italy-An Observational Study
Status: Completed | Type: Observational
Sponsor: Marco Marchetti (Other)
Collaborators: Azienda Ospedaliero Universitaria Maggiore della Carita (Other); Azienda Sanitaria Locale ASL 6, Livorno (Other Government); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Ospedale Civile - Padova (Unknown); S. Andrea Hospital (Other); Azienda Policlinico Umberto I (Other); San Carlo Public Hospital, Potenza, Italy (Other); Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other); Policlinico Universitario, Catania (Other); Azienda Ospedaliera Sant'Anna (Other); Ospedale di Cattinara - Azienda Universitaria Integrata -Trieste (Unknown); Abbott (Industry); Informapro Srl (Other)
Responsible Party: Sponsor-Investigator, Marco Marchetti, Director of the National Health Technology Assessment Centre, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Other Study IDs: TROCAR 2017
Record Dates: First submitted 2018-03-15; First posted 2018-04-05 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: NSTEMI - Non-ST Segment Elevation MI
Keywords: Troponin
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Myocardial infarction is one of the leading causes of death and disability worldwide. In addition to standard diagnostic methods, it has been shown that high-sensitivity cardiac troponin assays allow greater sensitivity in the diagnosis of myocardial infarction and assume a central role for both exclusion ("rule out") and confirmation ("rule in") of acute myocardial infarction , while allowing to reduce the time interval between ER admission and presumptive diagnosis.

Considering the relevance of this topic, we propose to conduct an observational study in real world clinical practice settings at Emergency Departments, aiming to evaluate clinical and economic aspects deriving from the use of the different quantitative assays of high-sensitivity cardiac troponin currently available in patients with suspected acute myocardial infarction and non-ST-elevation ECG (NSTEMI) on the admission, including time of diagnosis and number of laboratory and imaging tests performed.

DETAILED DESCRIPTION:
Observational, prospective, real-world clinical practice, multicentric study, conducted at 12 Emergency Departments in Italy.

Patients with suspected non-ST-elevation myocardial infarction (NSTEMI) who have undergone at least one high-sensitivity cardiac troponin test will be included.

Patients will be enrolled in the study after verification of selection criteria.

Enrollment is consecutive; each Center will suspend enrollment when it has reached the expected number of patients.

An electronic data collection form (eCRF) will be used to automatically generate an enrollment number to identify each patient.

Given the observational nature of the study, high-sensitivity cardiac troponin assays will be used according to current clinical practice.

Patients will be examined in the ED, and on a 30-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest pain
* Performing at least one cardiac troponin determination test
* Written informed consent

Exclusion Criteria:

* Refusal to provide informed consent
* Elevation of the ST segment to the ECG
* Pregnancy or breastfeeding
* Any other clinical condition not judged by the investigator compatible with participation in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the Emergency Department with chest pain
Sampling Method: Non-Probability Sample
Enrollment: 2913 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Time to diagnosis in the emergency department | 1-3-6 hours
  Time from admission at the emergency department and diagnosis or exclusion of NSTEMI

SECONDARY OUTCOMES:
Number of ruled-in and ruled-out patients | 1-3-6 hours
  Number of patients diagnosed with NSTEMI and hospitalized, and number of patients discharged from the emergency room after exclusion of NSTEMI
Number of tests performed | 1-3-6 hours
  Number of high-sensitivity cardiac troponin tests performed
Number of patients diagnosed with a Major Adverse Clinical Event | 30 days after the first assessment
  number of patients with myocardial infarction, stroke, or unplanned revascularization
30-day mortality | 30 days following admission
  Death rate 30 days after admission to the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Marco Marchetti, MD, Principal Investigator — Istituto Superiore di Sanità
Locations (1):
- Istituto Superiore di Sanità, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for Universal Definition of Myocardial Infarction; Authors/Task Force Members Chairpersons; Thygesen K, Alpert JS, White HD; Biomarker Subcommittee; Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA; ECG Subcommittee; Chaitman BR, Clemmensen PM, Johanson P, Hod H; Imaging Subcommittee; Underwood R, Bax JJ, Bonow JJ, Pinto F, Gibbons RJ; Classification Subcommittee; Fox KA, Atar D, Newby LK, Galvani M, Hamm CW; Intervention Subcommittee; Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J; Trials & Registries Subcommittee; Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML; Trials & Registries Subcommittee; Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G; Trials & Registries Subcommittee; Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D; Trials & Registries Subcommittee; Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG); Bax JJ, Baumgartner H, Ceconi C, Dean V, Deaton C, Fagard R, Funck-Brentano C, Hasdai D, Hoes A, Kirchhof P, Knuuti J, Kolh P, McDonagh T, Moulin C, Popescu BA, Reiner Z, Sechtem U, Sirnes PA, Tendera M, Torbicki A, Vahanian A, Windecker S; Document Reviewers; Morais J, Aguiar C, Almahmeed W, Arnar DO, Barili F, Bloch KD, Bolger AF, Botker HE, Bozkurt B, Bugiardini R, Cannon C, de Lemos J, Eberli FR, Escobar E, Hlatky M, James S, Kern KB, Moliterno DJ, Mueller C, Neskovic AN, Pieske BM, Schulman SP, Storey RF, Taubert KA, Vranckx P, Wagner DR. Third universal definition of myocardial infarction. J Am Coll Cardiol. 2012 Oct 16;60(16):1581-98. doi: 10.1016/j.jacc.2012.08.001. Epub 2012 Sep 5. No abstract available. PMID 22958960
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S. [2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC)]. G Ital Cardiol (Rome). 2016 Oct;17(10):831-872. doi: 10.1714/2464.25804. No abstract available. Italian. PMID 27869901
- [Background] Apple FS, Collinson PO; IFCC Task Force on Clinical Applications of Cardiac Biomarkers. Analytical characteristics of high-sensitivity cardiac troponin assays. Clin Chem. 2012 Jan;58(1):54-61. doi: 10.1373/clinchem.2011.165795. Epub 2011 Sep 30. PMID 21965555
- [Background] Apple FS, Ler R, Murakami MM. Determination of 19 cardiac troponin I and T assay 99th percentile values from a common presumably healthy population. Clin Chem. 2012 Nov;58(11):1574-81. doi: 10.1373/clinchem.2012.192716. Epub 2012 Sep 14. PMID 22983113
- [Background] Shah AS, Anand A, Sandoval Y, Lee KK, Smith SW, Adamson PD, Chapman AR, Langdon T, Sandeman D, Vaswani A, Strachan FE, Ferry A, Stirzaker AG, Reid A, Gray AJ, Collinson PO, McAllister DA, Apple FS, Newby DE, Mills NL; High-STEACS investigators. High-sensitivity cardiac troponin I at presentation in patients with suspected acute coronary syndrome: a cohort study. Lancet. 2015 Dec 19;386(10012):2481-8. doi: 10.1016/S0140-6736(15)00391-8. Epub 2015 Oct 8. PMID 26454362
- [Background] Rubini Gimenez M, Twerenbold R, Jaeger C, Schindler C, Puelacher C, Wildi K, Reichlin T, Haaf P, Merk S, Honegger U, Wagener M, Druey S, Schumacher C, Krivoshei L, Hillinger P, Herrmann T, Campodarve I, Rentsch K, Bassetti S, Osswald S, Mueller C. One-hour rule-in and rule-out of acute myocardial infarction using high-sensitivity cardiac troponin I. Am J Med. 2015 Aug;128(8):861-870.e4. doi: 10.1016/j.amjmed.2015.01.046. Epub 2015 Mar 31. PMID 25840034
- [Background] Shah AS, Griffiths M, Lee KK, McAllister DA, Hunter AL, Ferry AV, Cruikshank A, Reid A, Stoddart M, Strachan F, Walker S, Collinson PO, Apple FS, Gray AJ, Fox KA, Newby DE, Mills NL. High sensitivity cardiac troponin and the under-diagnosis of myocardial infarction in women: prospective cohort study. BMJ. 2015 Jan 21;350:g7873. doi: 10.1136/bmj.g7873. PMID 25609052
- [Background] Casagranda I, Cavazza M, Clerico A, Galvani M, Ottani F, Zaninotto M, Biasucci LM, Cervellin G, Lenzi T, Lippi G, Plebani M, Tubaro M. Proposal for the use in emergency departments of cardiac troponins measured with the latest generation methods in patients with suspected acute coronary syndrome without persistent ST-segment elevation. Clin Chem Lab Med. 2013 Sep;51(9):1727-37. doi: 10.1515/cclm-2013-0423. PMID 23893689
- [Background] Cremonesi P, Di Bella E, Montefiori M. Cost analysis of emergency department. J Prev Med Hyg. 2010 Dec;51(4):157-63. PMID 21553561
- [Background] Keller T, Zeller T, Ojeda F, Tzikas S, Lillpopp L, Sinning C, Wild P, Genth-Zotz S, Warnholtz A, Giannitsis E, Mockel M, Bickel C, Peetz D, Lackner K, Baldus S, Munzel T, Blankenberg S. Serial changes in highly sensitive troponin I assay and early diagnosis of myocardial infarction. JAMA. 2011 Dec 28;306(24):2684-93. doi: 10.1001/jama.2011.1896. PMID 22203537
- [Background] Reichlin T, Irfan A, Twerenbold R, Reiter M, Hochholzer W, Burkhalter H, Bassetti S, Steuer S, Winkler K, Peter F, Meissner J, Haaf P, Potocki M, Drexler B, Osswald S, Mueller C. Utility of absolute and relative changes in cardiac troponin concentrations in the early diagnosis of acute myocardial infarction. Circulation. 2011 Jul 12;124(2):136-45. doi: 10.1161/CIRCULATIONAHA.111.023937. Epub 2011 Jun 27. PMID 21709058
- [Background] Pickering JW, Greenslade JH, Cullen L, Flaws D, Parsonage W, George P, Worster A, Kavsak PA, Than MP. Validation of presentation and 3 h high-sensitivity troponin to rule-in and rule-out acute myocardial infarction. Heart. 2016 Aug 15;102(16):1270-8. doi: 10.1136/heartjnl-2015-308505. Epub 2016 Mar 8. PMID 26955848

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT03489603/SAP_000.pdf
  • Study Protocol (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT03489603/Prot_001.pdf